CLINICAL TRIAL: NCT04979910
Title: An Experimental Therapeutics Study of a Monoclonal Antibody Against Interleukin 17A in Patients With Treatment-Resistant Depression
Brief Title: Targeting IL-17A for Treatment-Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, James Murrough, Associate Professor of Psychiatry and Neuroscience, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 20-1909
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
Keywords: depression; investigational medication; treatment resistant depression; inflammation; ixekizumab; major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder, Treatment-Resistant; Inflammation | interventions — ixekizumab

STUDY DESIGN:
Intervention Model Description: This trial is a phase II, open-label trial where n=20 patients with treatment resistant depression will be treated with ixekizumab for 4 weeks and will undergo brain scans before and after the treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ixekizumab (Experimental): Ixekizumab 160 mg (two 80 mg injections) at Week 0, followed by 80 mg at Weeks 2 and 4 via subcutaneous route.
  Interventions: Drug: Ixekizumab

INTERVENTIONS:
Drug: Ixekizumab — a monoclonal antibody (mAb) against interleukin 17A (IL-17A)

SUMMARY:
The proposed study aims to test ixekizumab, a monoclonal antibody (mAb) against interleukin 17A (IL-17A), in patients with treatment-resistant depression (TRD).

DETAILED DESCRIPTION:
In the proposed study n=20 adult individuals with TRD will be treated with ixekizumab for 4 weeks. Participants will complete screening procedures, body fluid analyses and brain imaging before and after treatment with ixekizumab.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (and assent when applicable) obtained from subject;
* Ability for subject to comply with the requirements of the study as determined by the PI;
* Men and women, age 18-70 years;
* Participants must meet DSM-5 criteria for Major Depressive Disorder [MDD]) in a current major depressive episode (MDE) as determined by a study psychiatrist and confirmed using the Structured Clinical Interview for DSM-5 Research Version (SCID-5-RV);
* Participants have had ≥ 2 adequate trials of antidepressants/augmentation strategies during current episode. (Refer to ATRQ Guidelines for Completion for guidelines on dose/duration required for a trial to be considered adequate.);
* Patients must be on a stable dose of antidepressant medication for >4 weeks prior to randomization;
* Quick Inventory of Depressive Symptoms - Clinician Administered (QIDS-C) score ≥ 14
* If female of childbearing potential, must agree to use of a medically accepted form of contraception, or else agree to abstinence until 6 months after the last dose of study drug.
* Male patients, if heterosexually active with a partner who is female of childbearing potential, pregnant, or breastfeeding, must agree to barrier contraception for the treatment period and for at least 6 months after the last dose of study drug. Female partners of male participants must use at least one form of highly effective contraception starting at least one cycle prior to male patient study drug initiation until 6 months after the last dose of study drug.

Exclusion Criteria:

* A primary psychiatric diagnosis other than MDD as defined by DSM-5; [comorbid anxiety disorders (including agoraphobia, generalized anxiety disorder, social anxiety disorder and panic disorder) and posttraumatic stress disorder (PTSD) are allowed];
* Has a history of schizophrenia or other psychotic disorder, major depressive disorder with psychotic features, or bipolar I or II disorder;
* Diagnosis of a major neurocognitive disorder;
* Meets criteria for a moderate or severe substance use disorder within the past 6 months, with the exception of nicotine use disorder;
* The patient is pregnant or breastfeeding;
* Any contraindication to MRI or gadolinium including claustrophobia, any trauma or surgery which may have left magnetic material in the body, magnetic implants or pacemakers, inability to lie still for 1 hour or more, any known allergy to gadolinium;
* Positive urine toxicology screen for illicit drugs at the time of screening;
* Serious and imminent risk of self-harm or violence as determined by the PI;
* History of suicide attempt in the past 2 years or screening CSSRS Ideation Score >2 in the past month;
* Clinically significant abnormalities of laboratory tests or physical examination;
* Any unstable medical illnesses including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease); endocrinologic, neurologic (including history of severe head injury), immunologic, or hematologic disease;
* Presence of TB as assessed by Quantiferon Gold test at screening;
* Concomitant treatments with other biologics or other immune-suppressant agents; PRN use of NSAIDs is permissible;
* Female participants who are pregnant, breastfeeding, or may become pregnant, or unwilling to practice birth control during participation in the study or the 6 months following;
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James W Murrough, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ixekizumab
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ixekizumab
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.29 (17.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Dropped-out
Description: The safety and feasibility of using ixekizumab in patients with TRD will be assessed by the completion of treatment measured as the receipt of all three Ixekizumab injections (160 mg at week 0, 80 mg at weeks 2 and 4). Drop-out rates will be calculated.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ixekizumab
Number analyzed (Participants) | 7
Participants | 0

2. Primary Outcome: Number of Anticipated and Unanticipated Adverse Events
Description: The incidence and frequency of all anticipated and unanticipated serious and non-serious adverse events
Time Frame: 6 weeks
Measure: Number; unit: events
Arm/Group | Ixekizumab
Number analyzed (Participants) | 7
events | 8

3. Secondary Outcome: Change in Montgomery-Åsberg Depression Rating Scale Score - Response Rate
Description: Response rate at week 6 as compared to baseline, defined as >=50% MADRS total score improvement.
  The Montgomery-Åsberg Depression Rating Scale (MADARS) is a 10-item instrument used for the evaluation of depressive symptoms in adults and for the assessment of any changes to those symptoms. Each of the 10 items is rated on a scale of 0 to 6, with differing descriptors for each item. These individual item scores are added together to form a total score, which can range between 0 and 60 points. The MADRS provides a measure of the overall level of depression. Higher score indicates poorer health outcome.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixekizumab
Number analyzed (Participants) | 7
score on a scale
  Baseline | 28.57 (6.55)
  6 weeks | 23.86 (10.07)

4. Secondary Outcome: Change in Montgomery-Åsberg Depression Rating Scale Score - Remission Rate
Description: Remission rate at week 6 as compared to baseline, defined as MADRS total score of <=10..
  The Montgomery-Åsberg Depression Rating Scale (MADARS) is a 10-item instrument used for the evaluation of depressive symptoms in adults and for the assessment of any changes to those symptoms. Each of the 10 items is rated on a scale of 0 to 6, with differing descriptors for each item. These individual item scores are added together to form a total score, which can range between 0 and 60 points. The MADRS provides a measure of the overall level of depression. Higher score indicates poorer health outcome.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixekizumab
Number analyzed (Participants) | 7
score on a scale
  baseline | 28.57 (6.55)
  6 weeks | 23.86 (10.07)

5. Secondary Outcome: Change in Quick Inventory of Depressive Symptomatology, Self-Report [QIDS-SR] Score
Description: The Quick Inventory of Depressive Symptomatology, Self-Report (QIDS-SR) is a 16-item self-rated instrument designed to assess the severity of depressive symptoms. The 16 items cover the nine symptom domains of major depression and are rated on a scale of 0-3. Total score ranges from 0 to 27, with ranges of 0-5 (normal), 6-10 (mild), 11-15 (moderate), 16-20 (moderate to severe), and 21+ (severe). Higher score indicates poorer health outcome.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixekizumab
Number analyzed (Participants) | 7
score on a scale
  baseline | 13.57 (4.04)
  6 weeks | 11.57 (5.50)

6. Secondary Outcome: Change in Snaith-Hamilton Pleasure Scale (SHAPS)
Description: The Snaith-Hamilton Pleasure Scale (SHAPS) is a well-validated 14-item self-report questionnaire commonly used to assess anhedonia. Each item on the SHAPS is worded so that higher scores indicate greater pleasure capacity. A total score can be derived by summing the responses to each item. Items answered with "strongly agree" are coded as "1", while a "strongly disagree" response was assigned a score of "4." Total scores on the SHAPS can range from 14 to 56, with higher scores corresponding to higher levels of anhedonia.
Time Frame: Up to Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixekizumab
Number analyzed (Participants) | 7
score on a scale
  baseline | 35.29 (11.43)
  6 weeks | 33.14 (12.23)

7. Secondary Outcome: Change in Temporal Experience of Pleasure Scale
Description: The Temporal Experience of Pleasure Scale (TEPS) is an 18-item self-report measurement of anhedonia which consists of a series of statements that must be rated according to how accurate they are for the individual. The scale produces a sub-score that differentiates the role of anticipatory pleasure ('wanting') and is derived of 10 items. Subscales scores from 9-54. Total scores range is 16-108. Lower scores indicate greater levels of anhedonia.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixekizumab
Number analyzed (Participants) | 7
score on a scale
  baseline | 57.71 (21.78)
  6 weeks | 63.14 (24.59)

8. Secondary Outcome: Change in Clinical Global Impression Scale
Description: This is a widely administered clinician rated scale that assesses the subject overall illness severity and the degree of improvement from the initial assessment.
  Illness severity is rated on a 1-7 scale where 1 corresponds to "Normal, Not at All Ill", 2 is "Borderline Mentally Ill", the anchor for 3 is "Mildly Ill", the anchor for 4 is "Moderately Ill", 5 is "Markedly Ill", 6 is "Severely Ill", and 7 is "Among the Most Extremely Ill Patients". Illness improvement is rated on a 1-7 scale where 1 corresponds to "Very Much Improved", 2 is "Much Improved", the anchor for 3 is "Minimally Improved", the anchor for 4 is "No Change", 5 is "Minimally Worse", 6 is "Much Worse", and 7 is "Very Much Worse".
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixekizumab
Number analyzed (Participants) | 7
score on a scale
  Baseline CGI - Improvement | 3.43 (1.51)
  6 weeks - Improvement | 3.57 (0.98)
  baseline - Severity | 4.71 (0.49)
  6 weeks - Severity | 4.29 (0.76)

9. Secondary Outcome: Change in The Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) is a comprehensive, semi-structured interview that uniquely measures the full spectrum of suicidality including passive and active suicidal ideation, suicidal intent as well as suicidal behaviors. Full range from 0 to 9, with higher score indicating higher suicidal ideation severity.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixekizumab
Number analyzed (Participants) | 7
score on a scale
  Baseline | 0.86 (1.21)
  6 weeks | 0.57 (1.13)

10. Secondary Outcome: Change in The Hamilton Anxiety Rating Scale (HAM-A)
Description: The Hamilton Anxiety Rating Scale (HAM-A) is a scale of assessments of anxiety states. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Higher score indicates poorer health outcomes.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixekizumab
Number analyzed (Participants) | 7
score on a scale
  baseline | 19.00 (5.57)
  6 weeks | 14.86 (7.01)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Ixekizumab
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixekizumab (N=7)
Headache (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Tinnitus (Nervous system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Hot Flashes (Nervous system disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Palpitation (Cardiac disorders) | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT04979910/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT04979910/ICF_001.pdf